CLINICAL TRIAL: NCT04676828
Title: Functional Lung Avoidance SPECT-guided (ASPECT) Radiation Therapy for Lung Cancer Patients: Phase II Randomised Clinical Trial
Brief Title: Functional Lung Avoidance SPECT-guided Radiation Therapy of Lung Cancer
Acronym: ASPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Westmead and Blacktown Hospital, Sydney West Radiation Oncology Network, Sydney, Australia (Unknown); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Katherina Farr, MD, PhD, Specialist in Clinical Oncology, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFE-1930
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Radiation-Induced Disorder; Radiation Pneumonitis; Pulmonary Disease; Lung Function Decreased
Keywords: radiation-induced lung toxicity; functional avoidance methodology; radiation therapy of lung cancer
MeSH Terms: conditions — Lung Neoplasms; Abnormalities, Radiation-Induced; Radiation Pneumonitis; Lung Diseases; Respiratory Insufficiency | interventions — Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded phase 2
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers and outcome assessors are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPECT functional avoidance treatment (Experimental): SPECT-based radiation therapy given taken functional distribution in the lung into account, that avoids highly functional lung volumes sparing them from radiation.
  Interventions: Diagnostic Test: Single-photon-emission CT scan
- Standard treatment (No Intervention): CT-based radiation therapy given over 5- 6.5 weeks.

INTERVENTIONS:
Diagnostic Test: Single-photon-emission CT scan — SPECT/CT scan is an established functional modality used in the diagnosis and monitoring of lung disease. SPECT/CT scan images pulmonary circulation, where perfused areas equate with normal functional lung
  Arms: SPECT functional avoidance treatment

SUMMARY:
Study aims to determine if functional lung avoidance based on perfusion single photon emission (SPECT)/CT scan, improves toxicity outcomes for patients with advanced lung cancer undergoing chemo-radiotherapy. Functional avoidance implies a dose plan that takes functional distribution in the lung into account, and avoids highly functional lung volumes sparing them from radiation.

DETAILED DESCRIPTION:
In this project, a novel method of safe radiotherapy delivery shall be tested for patients with lung cancer in a clinical setting. Functional avoidance radiotherapy is a new method that protect highly functional lung tissue from radiation, while delivering high dose radiotherapy to the lung tumour. Radiotherapy is usually based on a CT scan that does not account for functional variations in the lungs. Therefore, I hypothesize that using functional distribution in the lungs and avoiding irradiation of highly functional lung will improve treatment outcome for individual patients with lung cancer.

The objective of my project is to determine if functional image guided radiotherapy (functional avoidance radiotherapy) improves toxicity outcomes for patients with lung cancer undergoing curative chemo-radiotherapy in a prospective clinical trial.

To reach this objective, the impact of functional avoidance radiotherapy on pulmonary toxicity measured by the incidence and severity of radiation-induced lung disease shall be assessed. Additionally, loco-regional control, time to progression, overall survival, quality of life and radiation-induced molecular response in patients treated with functional avoidance radiotherapy shall be assessed and compared to patients receiving standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified lung cancer (small-cell and non-small cell lung cancer)
* referred for radiotherapy with curative intent
* radiation dose of 60-66 Gy given in 2-Gy fractions, other dose levels and fractionation schedules accepted, as per site standard
* concurrent chemotherapy is accepted
* patients with oligometastatic disease are allowed, where metastasis have been ablated with surgery or radiotherapy
* receiving (chemo)-radiotherapy to the thoracic disease with curative intent
* adults over 18, that have given oral and written informed consent before patient registration.

Exclusion Criteria:

* concurrent immunotherapy
* previous radiotherapy to the thorax
* other uncontrolled malignancies; any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiation-induced lung toxicity | Measured serially from 1 to 12 months after treatment completion
  crude rate of symptomatic radiation-induced lung toxicity of grade 2 and higher. According to the Common Toxicity Criteria for Adverse Events version 5.0 for radiation pneumonitis, dyspnea, cough, or any other radiation-induced respiratory, thoracic and mediastinal disorder.

SECONDARY OUTCOMES:
Quality of life | Measured serially from 1 to 12 months after treatment completion
  Change in quality of life according to the European Organisation for Research and Treatment of Cancer quality of life questionnaires
Patient reported lung symptoms | Measured serially from 1 to 12 months after treatment completion
  Change in lung symptoms according to the European Organisation for Research and Treatment of Cancer questionnaire
Progression-free survival | at 12 months
  time from randomization to disease progression at any site or death
Overall survival | at 12 months
  time from randomization to death of any cause or last date known alive
Loco-regional control rate | at 12 months
  freedom from local disease progression

CONTACTS AND LOCATIONS:
Locations (2):
- Sydney West Radiation Oncology Network Westmead and Blacktown Hospitals, Sydney, New South Wales, Australia
- Department of Oncology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khalil AA, Hau E, Gebski V, Grau C, Gee H, Nyeng TB, West K, Kramer S, Farlow D, Knap M, Moller DS, Hoffmann L, Farr KP. Personal innovative approach in radiation therapy of lung cancer- functional lung avoidance SPECT-guided (ASPECT) radiation therapy: a study protocol for phase II randomised double-blind clinical trial. BMC Cancer. 2021 Aug 21;21(1):940. doi: 10.1186/s12885-021-08663-1. PMID 34418994